CLINICAL TRIAL: NCT02780154
Title: A Phase 1 Trial to Evaluate the Safety and Infectivity of Direct Venous Inoculation of Aseptic, Purified, Cryopreserved Plasmodium Falciparum (7G8 and NF54) Sporozoites in Non-immune Adults in Baltimore, USA
Brief Title: PfSPZ Challenge in Non-immune Adults in Baltimore, USA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14-0040; HHSN272201300022I
Record Dates: First submitted 2016-05-12; First posted 2016-05-23 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2017-04-05

CONDITIONS: Plasmodium Falciparum Infection
Keywords: 7G8 clone; NF54 strain; Non-immune; PCR; PfSPZ Challenge; Plasmodium falciparum; qPCR; Sporozoites
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- 1600 7G8 PfSPZ (Experimental): N= 7-9 participants will receive 1600 7G8 PfSPZ DVI in a volume of 500mcL
  Interventions: Biological: PfSPZ (7G8) Challenge
- 3200 7G8 PfSPZ (Experimental): N= 9 participants will receive 3200 7G8 PfSPZ DVI in a volume of 500mcL
  Interventions: Biological: PfSPZ (7G8) Challenge
- 3200 NF54 PfSPZ (Experimental): N= 5-6 participants will receive 3200 NF54 PfSPZ DVI in a volume of 500mcL
  Interventions: Biological: PfSPZ (NF54) Challenge
- 4800 7G8 PfSPZ (Experimental): N= 2-3 participants will receive 4800 7G8 PfSPZ DVI in a volume of 500mcL
  Interventions: Biological: PfSPZ (7G8) Challenge
- 800 7G8 PfSPZ (Experimental): N= 7-9 participants will receive 800 7G8 PfSPZ DVI in a volume of 500mcL
  Interventions: Biological: PfSPZ (7G8) Challenge

INTERVENTIONS:
Biological: PfSPZ (7G8) Challenge — PfSPZ (7G8) is a candidate vaccine, it consists of a suspension of purified, live-attenuated cryopreserved Pf sporozoites in a cryoprotectant.
  Arms: 1600 7G8 PfSPZ; 3200 7G8 PfSPZ; 4800 7G8 PfSPZ; 800 7G8 PfSPZ
Biological: PfSPZ (NF54) Challenge — PfSPZ (NF54) is a candidate vaccine, it consists of a suspension of purified, live-attenuated cryopreserved Pf sporozoites in a cryoprotectant.
  Arms: 3200 NF54 PfSPZ

SUMMARY:
This is a single center, randomized and controlled human study to optimize controlled human malaria infection (CHMI) administered by direct venous inoculation (DVI). 36 healthy adults aged between 18 and 45 years, will be randomized to one of five groups and will be inoculated with PfSPZ Challenge DVI. Participation duration is estimated to be 2 months, while the study duration is planned to be 4 months. The primary objective of this study is to assess the safety and reactogenicity of PfSPZ Challenge administered by DVI using 7G8 and NF54 P. falciparum strains.

DETAILED DESCRIPTION:
The proposed study is a single center, randomized and controlled human study to optimize controlled human malaria infection (CHMI) administered by direct venous inoculation (DVI). 30 to 36 participants will be randomized to one of five groups and will be inoculated with PfSPZ Challenge DVI. All participants recruited will be healthy adults aged between 18 and 45 years. The study duration is 4 months, participation duration is estimated to be 2 months. Safety and infectivity data will be collected for each study product and dose-level. Sera will be collected at baseline and at study day 29 for antibody assays. Participants, and clinical and laboratory investigators will be blinded to group allocation. The study primary endpoint will be reached at study day 29, at which time an interim study report will be generated. The investigators, the sponsor, the data and statistical analysis team, and Sanaria staff will meet in person or by teleconference on day 43 to review infection, pre-patent period, and adverse event results. These results will be made available to members of the International PfSPZ Consortium (I-PfSPZ-C) and if required, to regulatory authorities, including the FDA, to facilitate other PfSPZ Challenge CHMI studies with the appropriate disclaimers. Participants will be followed as outpatients for malaria diagnosis, treatment and follow-up to study day 57. Malaria positivity will be determined by qPCR diagnostics with microscopy as a backup. Participants who test positive for malaria and those who remain negative at study day 29 will be treated with oral atovaquone-proguanil. The primary objective of this study is to assess the safety and reactogenicity of PfSPZ Challenge administered by DVI using 7G8 and NF54 P. falciparum strains. Secondary objectives are to 1) assess the infectivity of four escalating doses of direct venous inoculation (DVI) of the 7G8 clone in comparison with an established dose (100% infective) DVI of the NF54 strain and 2) assess the time to malaria patency for escalating doses of the 7G8 clone compared to a single dose of the NF54 strain.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between the ages of 18 and 45 years, inclusive 2. Able and willing to participate for the duration of the study 3. Able and willing to provide written (not proxy) informed consent 4. Provides informed consent and correctly answers greater than or equal to 70% on the post consent quiz before any study procedures, and is available for all study visits -Note: Two attempts permitted 5. Females of childbearing potential must agree to practice highly effective contraception -Note: Contraception must be practiced from 30 days before the time of enrollment until at least 30 days following inoculation (such as double barrier methods (condoms plus foam or spermicide, diaphragm plus foam or spermicide), licensed intrauterine devices (IUDs), intravaginal or intra/transdermal or oral hormonal methods initiated at least 30 days before inoculation or challenge, documented surgical sterilization via tubal ligation the essure procedure or hysterectomy, abstinence or a vasectomized partner). The contraceptive method should remain unchanged throughout the required period 6. Is in good health, as determined by vital signs (heart rate, blood pressure, oral temperature); medical history; normal laboratory ranges listed in Appendix C; and a physical examination -Note: hemoglobin, white blood cell count, platelet count, glucose (random), serum alanine aminotransferase (ALT), serum creatinine, urine protein and urine blood 7. Agree not to travel to a malaria endemic region during study days 1-29 8. Willing to avoid non-study related blood donation from screening until 3 years (45) following P. falciparum challenge 9. Able to understand and comply with planned study procedures including daily outpatient follow-up visits beginning 5 days after inoculation

Exclusion Criteria:

1. Any history of malaria infection, or travel to a malaria endemic region within 3 months before planned date of CHMI 2. History of long-term residence (>5 years) in an area known to have significant transmission of P. falciparum 3. Positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B surface antigen (HBsAg) 4. Positive sickle cell screening test or known hemoglobinopathy 5. Current or recent (within the last four weeks) treatment with parenteral or oral corticosteroids (intranasal or inhaled steroids are acceptable), or other immunosuppressive agents, or chemotherapy 6. Screening laboratory values outside protocol-specified acceptable normal ranges as noted in Appendix C, except hematuria>1+ detected during menses for females. Note: For females who are menstruating, urinalysis frequently tests positive for blood and is not an indicator of poor health status or increased risk; other exceptions include ALT and creatinine below the lower limit of the reference range 7. Known hypersensitivity to components of PfSPZ Challenge, atovaquone-proguanil or artemether-lumefantrine 8. History of acute or chronic medical conditions including, but not limited to, disorders of the liver, kidney, lung, heart, nervous system, or other metabolic or autoimmune/inflammatory conditions 9. History of anaphylaxis or severe hypersensitivity reaction 10. Receipt of an investigational product on study days -31 to -1 or planned receipt of an investigational product on study days 1-57. 11. Any condition that, in the opinion of the investigator, would affect a participant's ability to understand or comply with the study protocol or would jeopardize a participant's safety or rights 12. Use or planned use of any drug with anti-malarial activity 30 days before or after CHMI Note: Medications with antimalarial activity include trimethoprim-sulfamethoxazole, azithromycin, erythromycin, tetracycline, doxycycline, minocycline, clindamycin, ciprofloxacin, levofloxacin, norfloxacin and rifampin 13. Planned surgery 30 days before or after CHMI 14. History of drug or alcohol abuse within the last five years 15. Receipt of blood or blood products in the previous six months or donation of a unit of blood within two months before screening 16. History of schizophrenia, bipolar disorder or other psychiatric condition that makes study compliance difficult Note: Subjects with psychoses or history of suicide attempt or gesture in the 3 years before study entry, ongoing risk for suicide. 17. History of diabetes mellitus with the exception of pregnancy-induced diabetes that has resolved 18. Has evidence of increased cardiovascular disease risk (defined as > 10%, 5 year risk) as determined by the method of Gaziano (46) Note: Risk factors include sex, age (years), systolic blood pressure (mm Hg), smoking status, body mass index (BMI, kg/mm2), reported diabetes status, and blood pressure. 19. Abnormal screening ECG Note: Pathologic Q wave and significant ST-T wave changes, left ventricular hypertrophy, non-sinus rhythm except isolated premature atrial or ventricular contractions, right of left bundle branch block, advanced A-V heart block (secondary or tertiary), QT/QTc interval >450 ms 20. Body mass index (BMI) >40 21. Known hypersensitivity to atovaquone-proguanil or artemether-lumefantrine 22. Anticipated medication use during the 28-day post-challenge period known to interact with atovaquone-proguanil or artemether-lumefantrine Note: Such as rifampin, carbamazepine, phenytoin, St. John's wort, cimetidine, metoclopramide, antacids, and kaolin 23. Personal beliefs that prevent receipt of human serum albumin 24. Immunization with more than three other vaccines within the past month and through study day 57 after CHMI 25. Previous vaccination with a candidate malaria vaccine or participation in a CHMI study 26. History of splenectomy 27. Pregnant or lactating females

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
The number and severity of local and systemic solicited and unsolicited reactogenicity symptoms related to PfSPZ Challenge for 7 days following DVI administration | Days 1-7
The number of serious adverse events recorded from study | Days 1-57

SECONDARY OUTCOMES:
Percent infectivity of each PfSPZ dose regimen | Days 1-57
Time to P. falciparum asexual parasitemia following experimental malaria challenge | Days 1-57

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland, United States